CLINICAL TRIAL: NCT01592526
Title: Autonomic Nervous Activity During the Systemic Inflammatory Response in Trained and Untrained Healthy Volunteers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Anders Rasmussen Rinnov, Local administrator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: H-3-2012-011
Record Dates: First submitted 2012-05-02; First posted 2012-05-07 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Systemic Inflammatory Response Syndrome
Keywords: Systemic inflammatory response.; Autonomic nervous regulation.; Cholinergic antiinflammatory pathway
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome | interventions — Endotoxins; Nicotine; Tobacco Use Cessation Devices; Nicotine Chewing Gum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Untrained, healthy volunteers A (Experimental): (Endotoxin) before (Endotoxin + Nicotine)
  Interventions: Other: Endotoxin; Other: Endotoxin + Nicotine
- Well-trained healthy volunteers A (Experimental): (Endotoxin) before (Endotoxin + Nicotine)
  Interventions: Other: Endotoxin; Other: Endotoxin + Nicotine
- Untrained, healthy volunteers B (Experimental): (Endotoxin + Nicotine) before (Endotoxin)
  Interventions: Other: Endotoxin; Other: Endotoxin + Nicotine
- Well-trained healthy volunteers B (Experimental): (Endotoxin + Nicotine) before (Endotoxin)
  Interventions: Other: Endotoxin; Other: Endotoxin + Nicotine

INTERVENTIONS:
Other: Endotoxin — Bolus injection of LPS 2 ng/kg IV at time = 2 hours (Study day A).
  Other Names: Clinical Center Reference Endotoxin
Other: Endotoxin + Nicotine — Transdermal application of nicotine patch applied at time = -8 hours (midnight the day before Study day B) + bolus injection of LPS 2 ng/kg at time = 2 hours (Study day 2)
  Other Names: Clinical Center Reference Endotoxin; Nicotine Patch (Nicorette 15mg/16t)

SUMMARY:
Critical illness, severe infection, extensive trauma or tissue damage cause an inflammatory (irritative) reaction in the body. This reaction affects the whole body and causes malaise, circulatory and cardiac changes, fever, increases the number of white blood cells in the blood stream and prompts release of signaling proteins. This reaction contributes to the development of considerable organ damage and possibly organ failure. These are serious complications in critical illness which are associated with a high mortality. This inflammatory reaction is affected by the autonomic nervous system. This is the part of the nervous system, which is beyond the control of the free will, and the part that regulates circulation, breathing and digestive functions. The autonomic nervous system works via so-called sympathetic signals, which set the body in a state of alertness to overcome immediate challenges, and parasympathetic (vagal) signals, which are especially active during restitution and rest. It is known, that the balanced activity in the autonomic nervous system affects the body's inflammatory response in critical illness. A study in mice has shown that if parasympathetic (vagal) signals are blocked mortality in critical illness is increased. Reversely, when the autonomic nervous system is medically stimulated towards parasympathetic signaling, the magnitude of the inflammatory response is decreased. Nicotine exerts this stimulatory effect.

Also, we know that individuals in good physical shape have increased parasympathetic tone compared to less trained individuals. However, studies have never addressed whether this shifted balance in the autonomic nervous system affects the inflammatory response related to critical illness.

Over the last 30 years an experimental model mimicking the inflammatory response has been used in studies. Inflammation may be simulated by injecting the drug E.Coli LPS, which induces a controlled, fully reversible, harmless reaction the duration of which is a few hours. Influenza-like symptoms occur and changes in circulatory parameters and concentrations of signaling proteins can be measured.

Using this experimental model, the investigators wish to study whether this shifted balance in the autonomic nervous system in individuals in good physical shape affects the body's reaction to critical illness. Investigators also want to determine how nicotine (using a nicotine patch) affects this reaction.

DETAILED DESCRIPTION:
Aim

The investigators wish to study the inflammatory response in very well-trained and relatively untrained healthy volunteers using the human endotoxemia model. Also, the investigators wish to study the effect on nicotine on the inflammatory response..

Background

1. Systemic inflammation and the endotoxin model

   Inflammation is the organisms response to invasion of microorganisms, trauma, endogenic or exogenic tissue damage. Systemic inflammation is a generalized response which affects the entire organism and presents with symptoms (malaise, shivering, dizziness, nausea), clinical manifestations (fever, tachypnea and hypocapnia, tachycardia) and biochemical findings such as altered numbers and relative composition of leucocytes in blood and increased concentrations of acute phase reactants and cytokines. Systemic inflammation, activated cascades and microcirculatory disruptions are considered important pathogenic elements ind the development of organ dysfunction, which is a frequent and serious complication to critical illness regardless of the underlying cause.

   Over the last 30 years the human endotoxemia model has been us as an experimental platform for studies of systemic inflammation. Since the year 1998 studies using this model have been conducted at Center for Inflammation and Metabolism (CIM), Rigshospitalet, Copenhagen University Hospital. An IV-bolus or infusion of E.Coli-lipopolysaccharide (LPS), an isolated component of the outer cell wall of Gram-negative bacteria, also referred to as endotoxin, is administered to healthy volunteers. A dose-dependent, fully reversible response is evoked the duration of which is a few hours with flu-like symptoms and production of pro- and anti-inflammatory markers, e.g tumor-necrosis-factor-α (TNF), interleukin(IL)-1β, IL-6, IL-1ra and IL-10. Serious adverse events have not been observed. The model is no accurate replication of acute infection, sepsis or other critical illness, however, evokes a reproducible, inter-individually comparable and fully reversible inflammatory response, which allows experimental studies of early stages of acute systemic inflammation and the interplay between different aspects of critical illness complicated by systemic inflammation.
2. The autonomic nervous system and the inflammatory response

   Activity in the autonomic nervous system affects the inflammatory response. Vagal stimulation inhibits release of pro-inflammatory cytokines, TNF-α, IL-1, IL-6 and high mobility group box protein-1 (HMGB-1), from macrophages activated by endotoxin, however, does not inhibit anti-inflammatory IL-10. Cytologic studies document, that this effect is mediated via the nicotinergic α7-subtype acetylcholine-receptor (α7nAchR). In a murine model peripheral vagal stimulation in vivo decreased mortality in endotoxemia and sepsis by cecal ligation.

   Kox et al found, that GTS-21 - a specific α7nAchR-agonist - was not generally associated with an altered inflammatory response in human endotoxemia, however, identified negative correlation between plasma concentrations of GTS-21 in the intervention group and maximal TNF-concentration.

   In another study, transdermally administered nicotine in healthy volunteers reduced the clinical, inflammatory response with reduced changes in body temperature and heart rate and increased plasma concentrations of cortisol and the anti-inflammatory IL-10. No differences in TNF-α, IL-1 or IL-6 expression were detected.
3. Heart rate variability

   Heart rate variability (HRV) is the variation in the interval between successive heart beats over time. It is a well-described phenomenon and is believed to reflect the cardiac balance of sympathetic- and vagal activity, thus changes in HRV may be interpreted as an indirect marker of changes in autonomic nervous activity. Physiological or pathological changes in autonomic nervous activity can be observed with performance of a standardized valsalva maneuver while monitoring blood pressure, heart rate and subsequent calculation of HRV and blood pressure variability.

   Reduced HRV is present in critical illness and is believed to reflect a shift in autonomic nervous balance towards increased sympathetic activity and vagal withdrawal. This phenomenon is a well documented predictor for poor outcome. Equally, reduced heart rate variability is observed in human endotoxemia in healthy volunteers. However, the magnitude of this reduction in HRV does not correspond to the severity of the inflammatory response as determined by plasma concentrations of pro-inflammatory cytokines.

   Individuals in excellent training status present altered activity in the autonomic nervous system with increased vagal activity with a low resting heart rate and increased HRV. Whether this altered autonomic activity still presents during critical illness is unknown, but it is a possibility that certain positive effects of physical activity may in part be due increased vagal activity and alterations in the systemic inflammatory response mediated by the vagal activity.
4. Exercise and the inflammatory response

No previous in vivo studies address the impact of increased vagal activity in well-trained individuals on the inflammatory response in comparison to that seen in untrained individuals. In the above mentioned study by Jan et al analysis of baseline HRV found that and HRV component traditionally considered proportional to sympathetic activity (LF/HF) correlated inversely with maximal TNF-α concentration in plasma. Furthermore, this study finds that heart rate at baseline does not correlate to HRV characteristics neither at baseline nor during endotoxemia. However, physical training condition of the participants is not reported.

Likewise, no mention of physical training status is made in the before mentioned studies concerning experimental use of nicotinergic agonist in endotoxemia (transdermally administered nicotine29 or orally administered GTS-21).

Two in vitro trials perform whole blood stimulation with LPS and find that baseline HRV is inversely proportional to TNF and IL-6 production, and inflammatory response in vitro is reduced in previously untrained individuals after a period of regular aerobic exercise. No in vivo studies addressing this have been conducted.

The investigators aim to study the inflammatory response in endotoxemia in well-trained and untrained healthy volunteers and determine whether transdermally administered nicotine alters this response.

A cross-over study design is applied so that volunteers act as their own control. This increases the chances of demonstrating a statistically significant effect.

Due to risk of LPS-tolerance the two study days need to be at least 4 weeks apart.

Hypotheses

1. Healthy well-trained individuals produce a reduced inflammatory response during experimental endotoxemia compared to untrained individuals.
2. Healthy, well-trained individuals display an increased HRV at baseline and experience a smaller reduction in HRV during endotoxemia compared to untrained individuals.
3. Transdermally administered nicotine during endotoxemia reduces clinical and preclinical features of the inflammatory response during endotoxemia in well-trained as well as untrained individuals.
4. Endotoxemia induces a transitory state of hyperalgesia in well-trained as well as untrained volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age 18-35 years
* BMI < 30 kg/m2
* Healthy
* Well-trained (N = 12): VO2max > 60 ml/kg/min
* Untrained (N = 12): VO2max < 47 ml/kg/min

Exclusion Criteria:

* Daily medicine intake (excl. antihistamines during pollen season)
* Smoking or use of nicotine substitutes
* Previous allergic reaction to nicotine pads
* Previous splenectomy

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2012-06; Primary Completion 2013-01 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Cytokines | up to 8 hours
  Cytokines are released into the bloodstream as part of the systemic inflammatory response and allow quantification of the severity of the systemic inflammatory response.
  Cytokines are measured multiple times to record changes from baseline during the intervention.

SECONDARY OUTCOMES:
Heart Rate Variability (HRV) | up to 8 hours
  HRV is the variation in the interval between heart beats over a given time period. A higher variability is considered an indirectly marker of increasing vagal acitivity. Low variability contrarily indicates decreasing vagal activity and increased sympathetic activity.
  HRV is calculated from continous, non-invasive monitoring of heart rhytm. Recordings are made at multiple fixed times to track changes from baseline during intervention.

OTHER OUTCOMES:
Pain Pressure Threshold (PPT) | Baseline, 2 hours, 6 hours
  Pressure algometry performed by a hand-held device with a tip area of 1 cm2 applied perpendicularly on the non-dominant lateral vastus muscle with a gradual increase in pressure until participant indicates painful stimuli.
Heat Pain Perception | Baseline, 2 hours, 6 hours
  A sequence of 4 tonic heat stimuli (45, 46, 47 and 48°C) delivered by a thermos with a duration of 5 s each and separated by an interstimulus interval of 30 s. Participants rated pain sensation using a visual analog scale (VAS).

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Janum, MD, Principal Investigator — Bispebjerg Hospital/Rigshospitalet; Kirsten Møller, MD,PhD,DMSc, Study Director — Rigshospitalet, Denmark
Locations (1):
- Center for Inflammation and Metabolism, Rigshospitalet, Copenhagen, Copenhagen OE, Denmark